CLINICAL TRIAL: NCT04925076
Title: Characterizing the Effects of Family History of Alcoholism on Alcohol Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB201800992-N; R01AA025337 (NIH)
Record Dates: First submitted 2021-06-08; First posted 2021-06-14 (Actual); Results first posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-07

CONDITIONS: Effects of Family History of Alcoholism and Sex on Alcohol Analgesia
Keywords: alcohol effects; pain
MeSH Terms: conditions — Pain | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: Participants will receive an active oral dose of alcohol or placebo in a counterbalanced manner.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family History Positive (Experimental): People reporting at least one parent with a history of alcohol problems.
  Interventions: Drug: Ethanol; Other: Placebo
- Family History Negative (Experimental): People who do not report having a parent with a history of alcohol problems.
  Interventions: Drug: Ethanol; Other: Placebo

INTERVENTIONS:
Drug: Ethanol — A beverage containing dose of ethanol individually determined to raise a participant's breath alcohol concentration up to approximately 0.08 g/dL.
Other: Placebo — A beverage that does not meaningfully increase breath alcohol concentration.

SUMMARY:
Self-medication of pain with alcohol is a common, yet risky, behavior. Evidence suggests family history of alcoholism may affect the degree to which alcohol use relieves pain, but the independent contributions of expectation and conditioning have not been previously studied. Interactive effects of sex and family history are also currently unclear. This project addresses this gap in knowledge and will inform further research and clinical/translational efforts for reducing risk associated with these behaviors.

ELIGIBILITY:
Inclusion Criteria:

- Consume at least 1 drink/month over the past 6 months

Exclusion Criteria:

* History of chronic pain
* Current use of opioids
* Current major depression
* History of any psychotic disorder
* Undercontrolled hypertension or diabetes
* History of neurologic disease
* History of serious medical illness
* History of drug or alcohol dependence, including nicotine, or a pattern of hazardous alcohol use
* Safety concerns related to MRI (for example, implants or pacing devices)

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 125 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Boissoneault, PhD, Principal Investigator — Assistant Professor
Locations (1):
- Center for Pain Research and Behavioral Health at UF Health, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Boissoneault J, Stennett B, Robinson ME. Acute alcohol intake alters resting state functional connectivity of nucleus accumbens with pain-related corticolimbic structures. Drug Alcohol Depend. 2020 Feb 1;207:107811. doi: 10.1016/j.drugalcdep.2019.107811. Epub 2019 Dec 24. PMID 31891860
- [Result] Sevel L, Stennett B, Schneider V 2nd, Bush N, Nixon SJ, Robinson M, Boissoneault J. Acute Alcohol Intake Produces Widespread Decreases in Cortical Resting Signal Variability in Healthy Social Drinkers. Alcohol Clin Exp Res. 2020 Jul;44(7):1410-1419. doi: 10.1111/acer.14381. Epub 2020 Jun 18. PMID 32472620

RESULTS

PARTICIPANT FLOW:
Groups:
- Family History Positive Men: Ethanol First, Then Placebo: Men with at least one parent with a history of alcohol problems, randomized to received ethanol first, followed by placebo. The first laboratory session lasted 4-8 hours, followed by a minimum 48 hour gap, and the second laboratory session lasted 4-8 hours. Ethanol: A beverage containing dose of ethanol individually determined to raise a participant's breath alcohol concentration up to approximately 0.08 g/dL. Placebo: A beverage that does not meaningfully increase breath alcohol concentration.
- Family History Negative Men: Ethanol First, Then Placebo: Men without a parent with a history of alcohol problems, randomized to received ethanol first, followed by placebo. The first laboratory session lasted 4-8 hours, followed by a minimum 48 hour gap, and the second laboratory session lasted 4-8 hours. Ethanol: A beverage containing dose of ethanol individually determined to raise a participant's breath alcohol concentration up to approximately 0.08 g/dL. Placebo: A beverage that does not meaningfully increase breath alcohol concentration.
- Family History Positive Men: Placebo First, Then Ethanol: Men with at least one parent with a history of alcohol problems, randomized to received placebo first, followed by ethanol. The first laboratory session lasted 4-8 hours, followed by a minimum 48 hour gap, and the second laboratory session lasted 4-8 hours. Ethanol: A beverage containing dose of ethanol individually determined to raise a participant's breath alcohol concentration up to approximately 0.08 g/dL. Placebo: A beverage that does not meaningfully increase breath alcohol concentration.
- Family History Negative Men: Placebo First, Then Ethanol: Men without a parent with a history of alcohol problems, randomized to received placebo first, followed by ethanol. The first laboratory session lasted 4-8 hours, followed by a minimum 48 hour gap, and the second laboratory session lasted 4-8 hours. Ethanol: A beverage containing dose of ethanol individually determined to raise a participant's breath alcohol concentration up to approximately 0.08 g/dL. Placebo: A beverage that does not meaningfully increase breath alcohol concentration.
- Family History Positive Women: Ethanol First, Then Placebo: Women with at least one parent with a history of alcohol problems, randomized to received ethanol first, followed by placebo. The first laboratory session lasted 4-8 hours, followed by a minimum 48 hour gap, and the second laboratory session lasted 4-8 hours. Ethanol: A beverage containing dose of ethanol individually determined to raise a participant's breath alcohol concentration up to approximately 0.08 g/dL. Placebo: A beverage that does not meaningfully increase breath alcohol concentration.
- Family History Negative Women: Ethanol First, Then Placebo: Women without a parent with a history of alcohol problems, randomized to received ethanol first, followed by placebo. The first laboratory session lasted 4-8 hours, followed by a minimum 48 hour gap, and the second laboratory session lasted 4-8 hours. Ethanol: A beverage containing dose of ethanol individually determined to raise a participant's breath alcohol concentration up to approximately 0.08 g/dL. Placebo: A beverage that does not meaningfully increase breath alcohol concentration.
- Family History Positive Women: Placebo First, Then Ethanol: Women with at least one parent with a history of alcohol problems, randomized to received placebo first, followed by ethanol. The first laboratory session lasted 4-8 hours, followed by a minimum 48 hour gap, and the second laboratory session lasted 4-8 hours. Ethanol: A beverage containing dose of ethanol individually determined to raise a participant's breath alcohol concentration up to approximately 0.08 g/dL. Placebo: A beverage that does not meaningfully increase breath alcohol concentration.
- Family History Negative Women: Placebo First, Then: Women without a parent with a history of alcohol problems, randomized to received placebo first, followed by ethanol. The first laboratory session lasted 4-8 hours, followed by a minimum 48 hour gap, and the second laboratory session lasted 4-8 hours. Ethanol: A beverage containing dose of ethanol individually determined to raise a participant's breath alcohol concentration up to approximately 0.08 g/dL. Placebo: A beverage that does not meaningfully increase breath alcohol concentration.
Period: Overall Study
Arm/Group | Family History Positive Men: Ethanol First, Then Placebo | Family History Negative Men: Ethanol First, Then Placebo | Family History Positive Men: Placebo First, Then Ethanol | Family History Negative Men: Placebo First, Then Ethanol | Family History Positive Women: Ethanol First, Then Placebo | Family History Negative Women: Ethanol First, Then Placebo | Family History Positive Women: Placebo First, Then Ethanol | Family History Negative Women: Placebo First, Then
Started | 10 | 17 | 12 | 14 | 12 | 23 | 18 | 19
Completed | 10 | 17 | 12 | 14 | 12 | 23 | 18 | 19
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Family History Positive Men: Men reporting at least one parent with a history of alcohol problems.
  Ethanol: A beverage containing dose of ethanol individually determined to raise a participant's breath alcohol concentration up to approximately 0.08 g/dL.
  Placebo: A beverage that does not meaningfully increase breath alcohol concentration.
- Family History Negative Men: Men who do not report having a parent with a history of alcohol problems.
  Ethanol: A beverage containing dose of ethanol individually determined to raise a participant's breath alcohol concentration up to approximately 0.08 g/dL.
  Placebo: A beverage that does not meaningfully increase breath alcohol concentration.
- Family History Positive Women: Women reporting at least one parent with a history of alcohol problems.
  Ethanol: A beverage containing dose of ethanol individually determined to raise a participant's breath alcohol concentration up to approximately 0.08 g/dL.
  Placebo: A beverage that does not meaningfully increase breath alcohol concentration.
- Family History Negative Women: Women who do not report having a parent with a history of alcohol problems.
  Ethanol: A beverage containing dose of ethanol individually determined to raise a participant's breath alcohol concentration up to approximately 0.08 g/dL.
  Placebo: A beverage that does not meaningfully increase breath alcohol concentration.
- Total: Total of all reporting groups
Arm/Group | Family History Positive Men | Family History Negative Men | Family History Positive Women | Family History Negative Women | Total
Number analyzed (Participants) | 22 | 31 | 30 | 42 | 125
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.09 (4.83) | 27.23 (5.64) | 25.13 (4.12) | 26.19 (4.40) | 25.75 (4.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 30 | 42 | 72
  Male | 22 | 31 | 0 | 0 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8 | 11 | 27
  Not Hispanic or Latino | 18 | 26 | 22 | 31 | 97
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 0 | 2
  Asian | 1 | 3 | 3 | 5 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 0 | 0 | 3
  White | 17 | 26 | 24 | 35 | 102
  More than one race | 1 | 1 | 2 | 2 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 22 | 31 | 30 | 42 | 125
Alcohol Use Disorders Identification Test [Mean (Standard Deviation); unit: total score] — The Alcohol Use Disorders Identification Test (AUDIT) is a standardized assessment of drinking frequency and heaviness, as well as consequences associated with alcohol intake. Higher scores reflect heavier/more frequent drinking and more severe alcohol-related consequences. Items are summed to compute total score, which can range from 0-40.
  total score | 4.45 (2.09) | 4.68 (1.45) | 4.70 (1.99) | 4.64 (1.61) | 4.63 (1.74)
Quantity-Frequency Index [Mean (Standard Deviation); unit: oz. absolute ethanol consumed per day] | .55 (.40) | .47 (.27) | .44 (.32) | .44 (.27) | .47 (.31)
Max Quantity [Mean (Standard Deviation); unit: oz. absolute ethanol] | 4.54 (2.66) | 5.05 (2.51) | 4.33 (2.50) | 4.16 (2.11) | 4.49 (2.41)
Expectancies for Alcohol Analgesia [Mean (Standard Deviation); unit: average score] — The Expectancies of Alcohol Analgesia questionnaire assesses perceived likelihood that using alcohol will reduce pain or improve pain coping. The EAA as administered consists of five 0-100 visual analog scales, which are averaged for analyses. Higher scores represent strong expectancies that alcohol is an effective analgesic.
  average score | 35.64 (26.20) | 44.46 (22.78) | 46.81 (19.40) | 42.53 (23.27) | 42.82 (22.68)

OUTCOME MEASURES:

1. Primary Outcome: Heat Pain Threshold
Description: Temperature of heat stimulus applied to the foot at which participant reports pain. VAS (visual analogue scale) pain intensity and unpleasantness ratings anchored from "no pain at all"/"not at all unpleasant" to "most intense/unpleasant imaginable" will be collected.
Time Frame: Day 1; Day 2 (Laboratory sessions will be separated by at least 48 hours.)
Measure: Mean (Standard Error); unit: degrees celsius
Arm/Group | Family History Positive Men | Family History Negative Men | Family History Positive Women | Family History Negative Women
Number analyzed (Participants) | 20 | 30 | 27 | 35
degrees celsius
  Alcohol Condition | 43.56 (.38) | 43.63 (.311) | 42.28 (.328) | 43.94 (.288)
  Placebo Condition | 43.20 (.386) | 43.43 (.315) | 41.98 (.33) | 43.75 (.29)
Statistical Analysis 1: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on pain threshold. Here we report the results of the analysis of the condition X family history X sex interaction; Test type: Superiority; p = .92, ANOVA; F(1,108)=.01
Statistical Analysis 2: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on pain threshold. Here we report the results of the analysis of the condition X sex interaction; Test type: Superiority; p = .92, ANOVA; F(1,108) = .01
Statistical Analysis 3: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on pain threshold. Here we report the results of the analysis of the condition X family history interaction; Test type: Superiority; p = .61, Chi-squared; F(1,108) = 0.27
Statistical Analysis 4: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on pain threshold. Here we report the results of the analysis of the family history X sex interaction; Test type: Superiority; p = .01, ANOVA; F(1,108) = 6.75
Statistical Analysis 5: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on pain threshold. Here we report the results of the analysis of the main effect of condition; Test type: Superiority; p = .05, ANOVA; F(1,108) = 3.83
Statistical Analysis 6: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on pain threshold. Here we report the results of the analysis of the main effect of family history; Test type: Superiority; p = .003, ANOVA; F(1,108) = 9.53
Statistical Analysis 7: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on pain threshold. Here we report the results of the analysis of the main effect of sex; Test type: Superiority; p = .12, ANOVA; F(1,108) = 2.41

2. Primary Outcome: Heat Pain Tolerance
Description: Temperature of heat stimulus applied to the foot at which participant no longer tolerates pain. VAS (visual analogue scale) pain intensity and unpleasantness ratings anchored from "no pain at all"/"not at all unpleasant" to "most intense/unpleasant imaginable" will be collected.
Time Frame: Day 1; Day 2 (Laboratory sessions will be separated by at least 48 hours.)
Measure: Mean (Standard Error); unit: degrees celsius
Arm/Group | Family History Positive Men | Family History Negative Men | Family History Positive Women | Family History Negative Women
Number analyzed (Participants) | 20 | 30 | 27 | 34
degrees celsius
  Alcohol Condition | 48.33 (.331) | 48.13 (.27) | 46.65 (.285) | 47.50 (.25)
  Placebo Condition | 48.18 (.339) | 47.95 (.277) | 46.57 (.29) | 47.68 (.257)
Statistical Analysis 1: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on pain tolerance. Here we report the results of the analysis of the condition X family history X sex interaction; Test type: Superiority; p = .38, ANOVA; F(1,107) = 0.78
Statistical Analysis 2: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on pain tolerance. Here we report the results of the analysis of the condition X sex interaction; Test type: Superiority; p = .27, ANOVA; F(1,107) = 0.27
Statistical Analysis 3: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on pain tolerance. Here we report the results of the analysis of the condition X family history interaction; Test type: Superiority; p = .70, ANOVA; F(1,107) = 0.15
Statistical Analysis 4: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on pain tolerance. Here we report the results of the analysis of the family history X sex interaction; Test type: Superiority; p = .05, ANOVA; F(1,107) = 3.87
Statistical Analysis 5: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on pain tolerance. Here we report the results of the analysis of the main effect of condition; Test type: Superiority; p = .03, ANOVA; F(1,107) = 5.18
Statistical Analysis 6: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on pain tolerance. Here we report the results of the analysis of the main effect of family history; Test type: Superiority; p = .14, ANOVA; F(1,107) = 2.24
Statistical Analysis 7: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on pain tolerance. Here we report the results of the analysis of the main effect of sex; Test type: Superiority; p < .001, ANOVA; F(1,107) = 17.25

3. Primary Outcome: Heat Pain Intensity Ratings
Description: Participant perception of pain at a temperature producing a pain rating of approximately 5 out of 10 at baseline. VAS (visual analogue scale) pain intensity ratings ranging from 0-100 and anchored from "no pain at all" to "most intense imaginable" will be collected. Higher values reflect ratings of more intense pain.
Time Frame: Day 1; Day 2 (Laboratory sessions will be separated by at least 48 hours.)
Measure: Mean (Standard Error); unit: units on a VAS
Arm/Group | Family History Positive Men | Family History Negative Men | Family History Positive Women | Family History Negative Women
Number analyzed (Participants) | 20 | 30 | 27 | 34
units on a VAS
  Alcohol Condition | 25.58 (3.43) | 25.48 (2.81) | 24.51 (2.98) | 27.11 (2.64)
  Placebo Condition | 28.41 (3.37) | 25.76 (2.75) | 24.07 (2.90) | 24.92 (2.58)
Statistical Analysis 1: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on pain intensity. Here we report the results of the analysis of the condition X family history X sex interaction; Test type: Superiority; p = .83, ANOVA; F(1,107) = 0.05
Statistical Analysis 2: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on pain intensity. Here we report the results of the analysis of the condition X sex interaction; Test type: Superiority; p = .12, ANOVA; F(1,107) = 2.43
Statistical Analysis 3: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on pain intensity. Here we report the results of the analysis of the condition X family history interaction; Test type: Superiority; p = .25, ANOVA; F(1,107) = 1.36
Statistical Analysis 4: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on pain intensity. Here we report the results of the analysis of the family history X sex interaction; Test type: Superiority; p = .58, ANOVA; F(1,107) = 0.31
Statistical Analysis 5: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on pain intensity. Here we report the results of the analysis of the main effect of condition; Test type: Superiority; p = .90, ANOVA; F(1,107) = 0.02
Statistical Analysis 6: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on pain intensity. Here we report the results of the analysis of the main effect of family history; Test type: Superiority; p = .95, ANOVA; F(1,107) = .004
Statistical Analysis 7: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on pain intensity. Here we report the results of the analysis of the main effect of sex; Test type: Superiority; p = .68, ANOVA; F(1,107) = 0.17

4. Primary Outcome: Perceived Pain Relief
Description: Rating of relief from pain associated with consumption of the study beverage. This is a VAS (visual analogue scale) assessing perceived pain relief ranging from 0-100 and anchored from "No relief at all" to "Most profound relief imaginable". Higher scores reflect greater perception of pain relief.
Time Frame: Day 1; Day 2 (Laboratory sessions will be separated by at least 48 hours.)
Measure: Mean (Standard Error); unit: units on a VAS
Arm/Group | Family History Positive Men | Family History Negative Men | Family History Positive Women | Family History Negative Women
Number analyzed (Participants) | 20 | 30 | 27 | 35
units on a VAS
  Alcohol Condition | 33.44 (4.41) | 32.18 (3.60) | 35.64 (3.78) | 37.60 (3.34)
  Placebo Condition | 13.63 (3.75) | 13.76 (3.06) | 14.83 (3.22) | 11.61 (2.83)
Statistical Analysis 1: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on pain relief. Here we report the results of the analysis of the condition X family history X sex interaction; Test type: Superiority; p = .36, ANOVA; F(1,107) = 0.83
Statistical Analysis 2: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on pain relief. Here we report the results of the analysis of the condition X sex interaction; Test type: Superiority; p = .24, ANOVA; F(1,108) = 1.41
Statistical Analysis 3: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on pain relief. Here we report the results of the analysis of the condition X family history interaction; Test type: Superiority; p = .60, ANOVA; F(1,108) = 0.28
Statistical Analysis 4: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on pain relief. Here we report the results of the analysis of the family history X sex interaction; Test type: Superiority; p = .99, ANOVA; F(1,108) = 0.00
Statistical Analysis 5: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on pain relief. Here we report the results of the analysis of the main effect of condition; Test type: Superiority; p < .001, ANOVA; F(1,108) = 139.63
Statistical Analysis 6: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on pain relief. Here we report the results of the analysis of the main effect of family history; Test type: Superiority; p = .84, ANOVA; F(1,108) = 0.04
Statistical Analysis 7: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on pain relief. Here we report the results of the analysis of the main effect of sex; Test type: Superiority; p = .59, ANOVA; F(1,108) = 0.30

5. Primary Outcome: Dorsolateral Prefrontal Cortex Activation
Description: Pain-related activation in the dorsolateral prefrontal cortex associated with application of painful heat vs. non-noxious warmth to the bottom of the right foot during fMRI acquisition. Scores are beta-weights associated with fit of activity within the region to activity predicted by convolving the canonical hemodynamic response function with the heat pain stimulus paradigm assessed using general linear modeling. Positive beta weights reflect activation associated with the stimulus paradigm, while negative beta weights reflect deactivation.
Time Frame: Day 1; Day 2 (Laboratory sessions will be separated by at least 48 hours.)
Measure: Mean (Standard Error); unit: beta weight
Arm/Group | Family History Positive Men | Family History Negative Men | Family History Positive Women | Family History Negative Women
Number analyzed (Participants) | 19 | 27 | 21 | 30
beta weight
  Alcohol Condition | -.01 (.054) | -.02 (.045) | .04 (.051) | .097 (.043)
  Placebo Condition | .099 (.047) | .019 (.039) | .082 (.044) | .115 (.037)
Statistical Analysis 1: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on dorsolateral prefrontal cortex activation. Here we report the results of the analysis of the condition X family history X sex interaction; Test type: Superiority; p = .66, ANOVA; F(1,93)=0.19
Statistical Analysis 2: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on dorsolateral prefrontal cortex activation. Here we report the results of the analysis of the condition X sex interaction; Test type: Superiority; p = .41, ANOVA; F(1,93)=0.69
Statistical Analysis 3: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on dorsolateral prefrontal cortex activation. Here we report the results of the analysis of the condition X family history interaction; Test type: Superiority; p = .39, ANOVA; F(1,93)=0.74
Statistical Analysis 4: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on dorsolateral prefrontal cortex activation. Here we report the results of the analysis of the family history X sex interaction; Test type: Superiority; p = .22, ANOVA; F(1,93)=1.54
Statistical Analysis 5: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on dorsolateral prefrontal cortex activation. Here we report the results of the analysis of the main effect of condition; Test type: Superiority; p = .06, ANOVA; F(1,93)=3.64
Statistical Analysis 6: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on dorsolateral prefrontal cortex activation. Here we report the results of the analysis of the main effect of family history; Test type: Superiority; p = .99, ANOVA; F(1,93)=0.000
Statistical Analysis 7: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on dorsolateral prefrontal cortex activation. Here we report the results of the analysis of the main effect of sex; Test type: Superiority; p = .09, ANOVA; F(1,93)=2.88

6. Primary Outcome: Hypothalamus Activation
Description: Pain-related activation in the hypothalamus associated with application of painful heat vs. non-noxious warmth to the bottom of the right foot during fMRI acquisition. Scores are beta-weights associated with fit of activity within the region to activity predicted by convolving the canonical hemodynamic response function with the heat pain stimulus paradigm assessed using general linear modeling. Positive beta weights reflect activation associated with the stimulus paradigm, while negative beta weights reflect deactivation.
Time Frame: Day 1; Day 2 (Laboratory sessions will be separated by at least 48 hours
Measure: Mean (Standard Error); unit: beta weight
Arm/Group | Family History Positive Men | Family History Negative Men | Family History Positive Women | Family History Negative Women
Number analyzed (Participants) | 19 | 27 | 21 | 30
beta weight
  Alcohol Condition | -.096 (.0449) | -.047 (.041) | .007 (.046) | -.036 (.039)
  Placebo Condition | -.083 (.047) | .018 (.04) | -.023 (.045) | -.022 (.038)
Statistical Analysis 1: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on hypothalamus activation. Here we report the results of the analysis of the condition X family history X sex interaction; Test type: Superiority; p = .55, ANOVA; F(1,93)=0.36
Statistical Analysis 2: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on hypothalamus activation. Here we report the results of the analysis of the condition X sex interaction; Test type: Superiority; p = .36, ANOVA; F(1,93)=0.84
Statistical Analysis 3: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on hypothalamus activation. Here we report the results of the analysis of the condition X family history interaction; Test type: Superiority; p = .36, ANOVA; F(1,93)=0.84
Statistical Analysis 4: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on hypothalamus activation. Here we report the results of the analysis of the family history X sex interaction; Test type: Superiority; p = .17, ANOVA; F(1,93)=1.93
Statistical Analysis 5: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on hypothalamus activation. Here we report the results of the analysis of the main effect of condition; Test type: Superiority; p = .55, ANOVA; F(1,93)=0.36
Statistical Analysis 6: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on hypothalamus activation. Here we report the results of the analysis of the main effect of family history; Test type: Superiority; p = .43, ANOVA; F(1,93)=0.63
Statistical Analysis 7: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; [analysis description as in outcome 1, analysis 7]; Test type: Superiority; p = .33, ANOVA; F(1,93)=0.96

7. Primary Outcome: Medial Prefrontal Cortex Activation
Description: Pain-related activation in the medial prefrontal cortex associated with application of painful heat vs. non-noxious warmth to the bottom of the right foot during fMRI acquisition. Scores are beta-weights associated with fit of activity within the region to activity predicted by convolving the canonical hemodynamic response function with the heat pain stimulus paradigm assessed using general linear modeling. Positive beta weights reflect activation associated with the stimulus paradigm, while negative beta weights reflect deactivation.
Time Frame: Day 1; Day 2 (Laboratory sessions will be separated by at least 48 hours.)
Measure: Mean (Standard Error); unit: beta weight
Arm/Group | Family History Positive Men | Family History Negative Men | Family History Positive Women | Family History Negative Women
Number analyzed (Participants) | 19 | 27 | 21 | 30
beta weight
  Alcohol Condition | -.173 (.081) | -.163 (.068) | -.096 (.077) | -.173 (.065)
  Placebo Condition | -.183 (.075) | -.201 (.063) | -.189 (.072) | -.15 (.06)
Statistical Analysis 1: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on medial prefrontal cortex activation. Here we report the results of the analysis of the condition X family history X sex interaction; Test type: Superiority; p = .34, ANOVA; F(1,93)=0.34
Statistical Analysis 2: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on medial prefrontal cortex activation. Here we report the results of the analysis of the condition X sex interaction; Test type: Superiority; p = .88, ANOVA; F(1,93)=0.02
Statistical Analysis 3: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on medial prefrontal cortex activation. Here we report the results of the analysis of the condition X family history interaction; Test type: Superiority; p = .56, ANOVA; F(1,93)=0.34
Statistical Analysis 4: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on medial prefrontal cortex activation. Here we report the results of the analysis of the family history X sex interaction; Test type: Superiority; p = .90, ANOVA; F(1,93)=0.02
Statistical Analysis 5: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on medial prefrontal cortex activation. Here we report the results of the analysis of the main effect of condition; Test type: Superiority; p = .45, ANOVA; F(1,93)=0.59
Statistical Analysis 6: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on medial prefrontal cortex activation. Here we report the results of the analysis of the main effect of family history; Test type: Superiority; p = .85, ANOVA; F(1,93)=0.04
Statistical Analysis 7: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on medial prefrontal cortex. Here we report the results of the analysis of the main effect of sex; Test type: Superiority; p = .64, ANOVA; F(1,93)=0.22

8. Primary Outcome: Nucleus Accumbens Activation
Description: Pain-related activation in the nucleus accumbens associated with application of painful heat vs. non-noxious warmth to the bottom of the right foot during fMRI acquisition. Scores are beta-weights associated with fit of activity within the region to activity predicted by convolving the canonical hemodynamic response function with the heat pain stimulus paradigm assessed using general linear modeling. Positive beta weights reflect activation associated with the stimulus paradigm, while negative beta weights reflect deactivation.
Time Frame: Day 1; Day 2 (Laboratory sessions will be separated by at least 48 hours.)
Measure: Mean (Standard Error); unit: beta weight
Arm/Group | Family History Positive Men | Family History Negative Men | Family History Positive Women | Family History Negative Women
Number analyzed (Participants) | 19 | 27 | 21 | 30
beta weight
  Alcohol Condition | -.037 (.041) | .055 (.034) | .075 (.039) | .131 (.033)
  Placebo Condition | .091 (.043) | .103 (.036) | .092 (.041) | .155 (.034)
Statistical Analysis 1: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on nucleus accumbens activation. Here we report the results of the analysis of the condition X family history X sex interaction; Test type: Superiority; p = .30, ANOVA; F(1,93)=1.07
Statistical Analysis 2: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on nucleus accumbens activation. Here we report the results of the analysis of the condition X sex interaction; Test type: Superiority; p = .11, ANOVA; F(1,93)=2.62
Statistical Analysis 3: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on nucleus accumbens activation. Here we report the results of the analysis of the condition X family history interaction; Test type: Superiority; p = .39, ANOVA; F(1,93)=0.76
Statistical Analysis 4: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on nucleus accumbens activation. Here we report the results of the analysis of the family history X sex interaction; Test type: Superiority; p = .89, ANOVA; F(1,93)=0.02
Statistical Analysis 5: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on nucleus accumbens activation. Here we report the results of the analysis of the main effect of condition; Test type: Superiority; p = .01, ANOVA; F(1,93)=6.72
Statistical Analysis 6: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on nucleus accumbens activation. Here we report the results of the analysis of the main effect of family history; Test type: Superiority; p = .08, ANOVA; F(1,93)=3.15
Statistical Analysis 7: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on nucleus accumbens activation. Here we report the results of the analysis of the main effect of sex; Test type: Superiority; p = .06, ANOVA; F(1,93)=3.71

9. Primary Outcome: Periaqueductal Gray Activation
Description: Pain-related activation in the periaqueductal gray associated with application of painful heat vs. non-noxious warmth to the bottom of the right foot during fMRI acquisition. Scores are beta-weights associated with fit of activity within the region to activity predicted by convolving the canonical hemodynamic response function with the heat pain stimulus paradigm assessed using general linear modeling. Positive beta weights reflect activation associated with the stimulus paradigm, while negative beta weights reflect deactivation.
Time Frame: Day 1; Day 2 (Laboratory sessions will be separated by at least 48 hours.)
Measure: Mean (Standard Error); unit: beta weight
Arm/Group | Family History Positive Men | Family History Negative Men | Family History Positive Women | Family History Negative Women
Number analyzed (Participants) | 19 | 27 | 21 | 30
beta weight
  Alcohol Condition | -.162 (.063) | -.089 (.053) | .055 (.060) | .052 (.05)
  Placebo Condition | .012 (.069) | -.038 (.058) | .036 (.066) | .059 (.055)
Statistical Analysis 1: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on periaqueductal gray activation. Here we report the results of the analysis of the condition X family history X sex interaction; Test type: Superiority; p = .29, ANOVA; F(1,93)=1.14
Statistical Analysis 2: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; [analysis description as in outcome 8, analysis 2]; Test type: Superiority; p = .10, ANOVA; F(1,93)=2.84
Statistical Analysis 3: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on periaqueductal gray activation. Here we report the results of the analysis of the condition X family history interaction; Test type: Superiority; p = .49, ANOVA; F(1,93)=0.47
Statistical Analysis 4: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on periaqueductal gray activation. Here we report the results of the analysis of the family history X sex interaction; Test type: Superiority; p = .99, ANOVA; F(1,93)=0.000
Statistical Analysis 5: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on periaqueductal gray activation. Here we report the results of the analysis of the main effect of condition; Test type: Superiority; p = .13, ANOVA; F(1,93)=2.29
Statistical Analysis 6: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on periaqueductal gray activation. Here we report the results of the analysis of the main effect of family history; Test type: Superiority; p = .82, ANOVA; F(1,93)=0.05
Statistical Analysis 7: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on periaqueductal gray activation. Here we report the results of the analysis of the main effect of sex; Test type: Superiority; p = 0.02, ANOVA; F(1,93)=6.09

10. Primary Outcome: Anterior Cingulate Cortex Activation
Description: Pain-related activation in the anterior cingulate cortex associated with application of painful heat vs. non-noxious warmth to the bottom of the right foot during fMRI acquisition. Scores are beta-weights associated with fit of activity within the region to activity predicted by convolving the canonical hemodynamic response function with the heat pain stimulus paradigm assessed using general linear modeling. Positive beta weights reflect activation associated with the stimulus paradigm, while negative beta weights reflect deactivation.
Time Frame: Day 1; Day 2 (Laboratory sessions will be separated by at least 48 hours.)
Measure: Mean (Standard Error); unit: beta weight
Arm/Group | Family History Positive Men | Family History Negative Men | Family History Positive Women | Family History Negative Women
Number analyzed (Participants) | 19 | 27 | 21 | 30
beta weight
  Alcohol Condition | .020 (.046) | .045 (.038) | .082 (.044) | .040 (.037)
  Placebo Condition | .049 (.044) | .038 (.037) | .066 (.042) | .080 (.035)
Statistical Analysis 1: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on anterior cingulate cortex activation. Here we report the results of the analysis of the condition X family history X sex interaction; Test type: Superiority; p = .32, ANOVA; F(1,93)=1.01
Statistical Analysis 2: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on anterior cingulate cortex activation. Here we report the results of the analysis of the condition X sex interaction; Test type: Superiority; p = .99, ANOVA; F(1,93)=0.000
Statistical Analysis 3: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on anterior cingulate cortex activation. Here we report the results of the analysis of the condition X family history interaction; Test type: Superiority; p = .83, ANOVA; F(1,93)=0.05
Statistical Analysis 4: Comparison: Family History Positive Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on anterior cingulate cortex activation. Here we report the results of the analysis of the family history X sex interaction; Test type: Superiority; p = .75, ANOVA; F(1,93)=0.10
Statistical Analysis 5: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on anterior cingulate cortex activation. Here we report the results of the analysis of the main effect of condition; Test type: Superiority; p = .62, ANOVA; F(1,93)=0.25
Statistical Analysis 6: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on anterior cingulate cortex activation. Here we report the results of the analysis of the main effect of family history; Test type: Superiority; p = .92, ANOVA; F(1,93)=0.01
Statistical Analysis 7: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on anterior cingulate cortex activation. Here we report the results of the analysis of the main effect of sex; Test type: Superiority; p = .39, ANOVA; F(1,93)=0.76

11. Primary Outcome: Amgydala Activation
Description: Pain-related activation in the amygdala associated with application of painful heat vs. non-noxious warmth to the bottom of the right foot during fMRI acquisition. Scores are beta-weights associated with fit of activity within the region to activity predicted by convolving the canonical hemodynamic response function with the heat pain stimulus paradigm assessed using general linear modeling. Positive beta weights reflect activation associated with the stimulus paradigm, while negative beta weights reflect deactivation.
Time Frame: Day 1; Day 2 (Laboratory sessions will be separated by at least 48 hours.)
Measure: Mean (Standard Error); unit: beta weight
Arm/Group | Family History Positive Men | Family History Negative Men | Family History Positive Women | Family History Negative Women
Number analyzed (Participants) | 19 | 27 | 21 | 30
beta weight
  Alcohol Condition | -.155 (.055) | -.039 (.046) | .013 (.052) | -.061 (.044)
  Placebo Condition | -.050 (.048) | -.007 (.040) | .011 (.046) | -.054 (.038)
Statistical Analysis 1: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on amygdala activation. Here we report the results of the analysis of the condition X family history X sex interaction; Test type: Superiority; p = .50, ANOVA; F(1,93)=0.45
Statistical Analysis 2: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on amygdala activation. Here we report the results of the analysis of the condition X sex interaction; Test type: Superiority; p = .28, ANOVA; F(1,93)=1.20
Statistical Analysis 3: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on amygdala activation. Here we report the results of the analysis of the condition X family history interaction; Test type: Superiority; p = .60, ANOVA; F(1,93)=0.28
Statistical Analysis 4: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on amygdala activation. Here we report the results of the analysis of the family history X sex interaction; Test type: Superiority; p = .04, ANOVA; F(1,93)=4.48
Statistical Analysis 5: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on amygdala activation. Here we report the results of the analysis of the main effect of condition; Test type: Superiority; p = .25, ANOVA; F(1,93)=1.37
Statistical Analysis 6: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on amygdala activation. Here we report the results of the analysis of the main effect of family history; Test type: Superiority; p = .89, ANOVA; F(1,93)=0.01
Statistical Analysis 7: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on amygdala activation. Here we report the results of the analysis of the main effect of sex; Test type: Superiority; p = .26, ANOVA; F(1,93)=1.28

12. Primary Outcome: Hippocampus Activation
Description: Pain-related activation in the hippocampus associated with application of painful heat vs. non-noxious warmth to the bottom of the right foot during fMRI acquisition. Scores are beta-weights associated with fit of activity within the region to activity predicted by convolving the canonical hemodynamic response function with the heat pain stimulus paradigm assessed using general linear modeling. Positive beta weights reflect activation associated with the stimulus paradigm, while negative beta weights reflect deactivation.
Time Frame: Day 1; Day 2 (Laboratory sessions will be separated by at least 48 hours.)
Measure: Mean (Standard Error); unit: beta weight
Arm/Group | Family History Positive Men | Family History Negative Men | Family History Positive Women | Family History Negative Women
Number analyzed (Participants) | 19 | 27 | 21 | 30
beta weight
  Alcohol Condition | -.154 (.048) | -.130 (.041) | -.116 (.046) | -.128 (.039)
  Placebo Condition | -.074 (.046) | -.083 (.039) | -.145 (.044) | -.158 (.037)
Statistical Analysis 1: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on hippocampus activation. Here we report the results of the analysis of the condition X family history X sex interaction; Test type: Superiority; p = .76, ANOVA; F(1,93)=0.09
Statistical Analysis 2: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on hippocampus activation. Here we report the results of the analysis of the condition X sex interaction; Test type: Superiority; p = .09, ANOVA; F(1,93)=3.00
Statistical Analysis 3: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on hippocampus activation. Here we report the results of the analysis of the condition X family history interaction; Test type: Superiority; p = .76, ANOVA; F(1,93)=0.10
Statistical Analysis 4: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on hippocampus activation. Here we report the results of the analysis of the family history X sex interaction; Test type: Superiority; p = .77, ANOVA; F(1,93)=0.09
Statistical Analysis 5: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on hippocampus activation. Here we report the results of the analysis of the main effect of condition; Test type: Superiority; p = .52, ANOVA; F(1,93)=0.41
Statistical Analysis 6: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on pain hippocampus activation. Here we report the results of the analysis of the main effect of family history; Test type: Superiority; p = .93, ANOVA; F(1,93)=0.007
Statistical Analysis 7: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on hippocampus activation. Here we report the results of the analysis of the main effect of sex; Test type: Superiority; p = .42, ANOVA; F(1,93)=0.64

13. Primary Outcome: Insula Activation
Description: Pain-related activation in the insula associated with application of painful heat vs. non-noxious warmth to the bottom of the right foot during fMRI acquisition. Scores are beta-weights associated with fit of activity within the region to activity predicted by convolving the canonical hemodynamic response function with the heat pain stimulus paradigm assessed using general linear modeling. Positive beta weights reflect activation associated with the stimulus paradigm, while negative beta weights reflect deactivation.
Time Frame: Day 1; Day 2 (Laboratory sessions will be separated by at least 48 hours.)
Measure: Mean (Standard Error); unit: beta weight
Arm/Group | Family History Positive Men | Family History Negative Men | Family History Positive Women | Family History Negative Women
Number analyzed (Participants) | 19 | 27 | 21 | 30
beta weight
  Alcohol Condition | .220 (.054) | .286 (.045) | .270 (.051) | .318 (.043)
  Placebo Condition | .389 (.055) | .298 (.046) | .329 (.052) | .312 (.044)
Statistical Analysis 1: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on insula activation. Here we report the results of the analysis of the condition X family history X sex interaction; Test type: Superiority; p = .44, ANOVA; F(1,93)=0.62
Statistical Analysis 2: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on insula activation. Here we report the results of the analysis of the condition X sex interaction; Test type: Superiority; p = .27, ANOVA; F(1,93)=1.23
Statistical Analysis 3: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on insula activation. Here we report the results of the analysis of the condition X family history interaction; Test type: Superiority; p = .06, ANOVA; F(1,93)=3.66
Statistical Analysis 4: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on insula activation. Here we report the results of the analysis of the family history X sex interaction; Test type: Superiority; p = .73, ANOVA; F(1,93)=0.13
Statistical Analysis 5: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on insula activation. Here we report the results of the analysis of the main effect of condition; Test type: Superiority; p = .047, ANOVA; F(1,93)=4.04
Statistical Analysis 6: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on insula activation. Here we report the results of the analysis of the main effect of family history; Test type: Superiority; p = .97, ANOVA; F(1,93)=0.001
Statistical Analysis 7: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on insula activation. Here we report the results of the analysis of the main effect of sex; Test type: Superiority; p = .82, ANOVA; F(1,93)=0.05

14. Primary Outcome: Postcentral Gyrus Activation
Description: Pain-related activation in the postcentral gyrus associated with application of painful heat vs. non-noxious warmth to the bottom of the right foot during fMRI acquisition. Scores are beta-weights associated with fit of activity within the region to activity predicted by convolving the canonical hemodynamic response function with the heat pain stimulus paradigm assessed using general linear modeling. Positive beta weights reflect activation associated with the stimulus paradigm, while negative beta weights reflect deactivation.
Time Frame: Day 1; Day 2 (Laboratory sessions will be separated by at least 48 hours.)
Measure: Mean (Standard Error); unit: beta weight
Arm/Group | Family History Positive Men | Family History Negative Men | Family History Positive Women | Family History Negative Women
Number analyzed (Participants) | 19 | 27 | 21 | 30
beta weight
  Alcohol Condition | -.139 (.046) | -.038 (.039) | -.068 (.044) | -.041 (.37)
  Placebo Condition | -.053 (.048) | -.085 (.041) | -.048 (.046) | -.077 (.039)
Statistical Analysis 1: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on postcentral gyrus activation. Here we report the results of the analysis of the condition X family history X sex interaction; Test type: Superiority; p = 0.45, ANOVA; F(1,93)=0.57
Statistical Analysis 2: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on postcentral gyrus activation. Here we report the results of the analysis of the condition X sex interaction; Test type: Superiority; p = .59, ANOVA; F(1,93)=0.29
Statistical Analysis 3: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on postcentral gyrus activation. Here we report the results of the analysis of the condition X family history interaction; Test type: Superiority; p = .07, ANOVA; F(1,93)=3.41
Statistical Analysis 4: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on postcentral gyrus activation. Here we report the results of the analysis of the family history X sex interaction; Test type: Superiority; p = .61, ANOVA; F(1,93)=0.26
Statistical Analysis 5: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on postcentral gyrus activation. Here we report the results of the analysis of the main effect of condition; Test type: Superiority; p = .82, ANOVA; F(1,93)=0.05
Statistical Analysis 6: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on postcentral gyrus activation. Here we report the results of the analysis of the main effect of family history; Test type: Superiority; p = .63, ANOVA; F(1,93)=0.23
Statistical Analysis 7: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on postcentral gyrus activation. Here we report the results of the analysis of the main effect of sex; Test type: Superiority; p = .55, ANOVA; F(1,93)=0.36

15. Primary Outcome: Thalamus Activation
Description: Pain-related activation in the thalamus associated with application of painful heat vs. non-noxious warmth to the bottom of the right foot during fMRI acquisition. Scores are beta-weights associated with fit of activity within the region to activity predicted by convolving the canonical hemodynamic response function with the heat pain stimulus paradigm assessed using general linear modeling. Positive beta weights reflect activation associated with the stimulus paradigm, while negative beta weights reflect deactivation.
Time Frame: Day 1; Day 2 (Laboratory sessions will be separated by at least 48 hours.)
Measure: Mean (Standard Error); unit: beta weight
Arm/Group | Family History Positive Men | Family History Negative Men | Family History Positive Women | Family History Negative Women
Number analyzed (Participants) | 19 | 27 | 21 | 30
beta weight
  Alcohol Condition | -.141 (.059) | -.076 (.049) | .023 (.056) | -.022 (.047)
  Placebo Condition | -.033 (.053) | -.027 (.044) | .066 (.050) | -.029 (.042)
Statistical Analysis 1: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on thalamus activation. Here we report the results of the analysis of the condition X family history X sex interaction; Test type: Superiority; p = .57, ANOVA; F(1,93)=0.32
Statistical Analysis 2: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on thalamus activation. Here we report the results of the analysis of the condition X sex interaction; Test type: Superiority; p = .14, ANOVA; F(1,93)=2.17
Statistical Analysis 3: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on thalamus activation. Here we report the results of the analysis of the condition X family history interaction; Test type: Superiority; p = .69, ANOVA; F(1,93)=0.32
Statistical Analysis 4: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on thalamus activation. Here we report the results of the analysis of the family history X sex interaction; Test type: Superiority; p = .34, ANOVA; F(1,93)=0.92
Statistical Analysis 5: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on thalamus activation. Here we report the results of the analysis of the main effect of condition; Test type: Superiority; p = 0.29, ANOVA; F(1,93)=1.16
Statistical Analysis 6: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on thalamus activation. Here we report the results of the analysis of the main effect of family history; Test type: Superiority; p = .95, ANOVA; F(1,93)=0.004
Statistical Analysis 7: Comparison: Family History Positive Men vs Family History Negative Men vs Family History Positive Women vs Family History Negative Women; 2 (beverage condition: alcohol vs. placebo) X 2 (family history: positive vs. negative) X 2 (sex: men vs. women) mixed general linear model on thalamus activation. Here we report the results of the analysis of the main effect of sex; Test type: Superiority; p = .11, ANOVA; F(1,93)=2.65

ADVERSE EVENTS:
Time Frame: Duration of study participation (4-8 hours per study session, with at least 48 hours separating each session)
Groups:
- Family History Positive Men - Alcohol Condition: Men reporting at least one parent with a history of alcohol problems who received a beverage containing alcohol (ethanol) during the laboratory session.
  Ethanol: A beverage containing dose of ethanol individually determined to raise a participant's breath alcohol concentration up to approximately 0.08 g/dL.
  Placebo: A beverage that does not meaningfully increase breath alcohol concentration.
- Family History Negative Men - Alcohol Condition: Men who do not report having a parent with a history of alcohol problems who received a beverage containing alcohol (ethanol) during the laboratory session.
  Ethanol: A beverage containing dose of ethanol individually determined to raise a participant's breath alcohol concentration up to approximately 0.08 g/dL.
  Placebo: A beverage that does not meaningfully increase breath alcohol concentration.
- Family History Positive Women - Alcohol Condition: Women reporting at least one parent with a history of alcohol problems who received a beverage containing alcohol (ethanol) during the laboratory session.
  Ethanol: A beverage containing dose of ethanol individually determined to raise a participant's breath alcohol concentration up to approximately 0.08 g/dL.
  Placebo: A beverage that does not meaningfully increase breath alcohol concentration.
- Family History Negative Women - Alcohol Condition: Women who do not report having a parent with a history of alcohol problems who received a beverage containing alcohol (ethanol) during the laboratory session.
  Ethanol: A beverage containing dose of ethanol individually determined to raise a participant's breath alcohol concentration up to approximately 0.08 g/dL.
  Placebo: A beverage that does not meaningfully increase breath alcohol concentration.
- Family History Positive Men - Placebo Condition: Men reporting at least one parent with a history of alcohol problems who received a placebo beverage during the laboratory session.
  Ethanol: A beverage containing dose of ethanol individually determined to raise a participant's breath alcohol concentration up to approximately 0.08 g/dL.
  Placebo: A beverage that does not meaningfully increase breath alcohol concentration.
- Family History Negative Men - Placebo Condition: Men who do not report having a parent with a history of alcohol problems who received a placebo beverage during the laboratory session.
  Ethanol: A beverage containing dose of ethanol individually determined to raise a participant's breath alcohol concentration up to approximately 0.08 g/dL.
  Placebo: A beverage that does not meaningfully increase breath alcohol concentration.
- Family History Positive Women - Placebo Condition: Women reporting at least one parent with a history of alcohol problems who received a placebo beverage during the laboratory session.
  Ethanol: A beverage containing dose of ethanol individually determined to raise a participant's breath alcohol concentration up to approximately 0.08 g/dL.
  Placebo: A beverage that does not meaningfully increase breath alcohol concentration.
- Family History Negative Women - Placebo Condition: Women who do not report having a parent with a history of alcohol problems who received a placebo beverage during the laboratory session.
  Ethanol: A beverage containing dose of ethanol individually determined to raise a participant's breath alcohol concentration up to approximately 0.08 g/dL.
  Placebo: A beverage that does not meaningfully increase breath alcohol concentration.
Arm/Group | Family History Positive Men - Alcohol Condition | Family History Negative Men - Alcohol Condition | Family History Positive Women - Alcohol Condition | Family History Negative Women - Alcohol Condition | Family History Positive Men - Placebo Condition | Family History Negative Men - Placebo Condition | Family History Positive Women - Placebo Condition | Family History Negative Women - Placebo Condition
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/31 | 0/30 | 0/42 | 0/22 | 0/31 | 0/30 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/31 | 0/30 | 0/42 | 0/22 | 0/31 | 0/30 | 0/42
Other Adverse Events (participants affected / at risk) | 0/22 | 0/31 | 0/30 | 0/42 | 0/22 | 0/31 | 0/30 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-04-05): https://cdn.clinicaltrials.gov/large-docs/76/NCT04925076/Prot_SAP_ICF_000.pdf